CLINICAL TRIAL: NCT01777750
Title: Strategic Target Temperature Management in Myocardial Infarction
Brief Title: Cooling in Myocardial Infarction
Acronym: STATIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Austrian Science Fund (FWF) (Other)
Responsible Party: Principal Investigator, Dr. Christoph Testori, Department of Emergency Medicine, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KLI209
Record Dates: First submitted 2013-01-23; First posted 2013-01-29 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2017-03

CONDITIONS: ST-elevation Myocardial Infarction
Keywords: Myocardial Infarction; Myocardial Reperfusion Injury; Reperfusion Injury; Anterior Wall Myocardial Infarction; Inferior Wall Myocardial Infarction; Pathologic Processes; Myocardial Ischemia
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction; Myocardial Reperfusion Injury; Reperfusion Injury; Anterior Wall Myocardial Infarction; Inferior Wall Myocardial Infarction; Pathologic Processes; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre- and perinterventional hypothermia (Active Comparator): Cooling will be initiated by the application of cooling pads in the out-of-hospital setting followed by an infusion of 1000-2000ml of cold saline. In the cath lab a endovascular cooling catheter will be placed into the inferior vena cava via a femoral vein to achieve a core temperature of <35°C prior to revascularization.
  Interventions: Device: EMCOOLS flex pad; Philips Innercool RTx
- Standard treatment (No Intervention): Standard treatment

INTERVENTIONS:
Device: EMCOOLS flex pad; Philips Innercool RTx — Surface cooling with EMCOOLS flex pads (out-of-hospital); Infusion of 1000ml to 2000ml of cold saline (out-of-hospital); central-venous cooling (Philips Inntercool RTx)
  Arms: Pre- and perinterventional hypothermia

SUMMARY:
The primary goal in the treatment of acute myocardial infarction is to reperfuse the ischemic myocardium to reduce infarct size. Animal data and human data suggest that whole-body cooling to temperatures below 35°C before revascularisation can additionally reduce infarct size and therefore improves outcome in these patients.

The purpose of the study is to determine if a combined cooling strategy started in the out-of-hospital arena is able to reduce infarct size in acute myocardial infarction.

DETAILED DESCRIPTION:
Background: Contemporary therapy in patients with an on-going ST-elevation myocardial infarction (STEMI) is to reperfuse the ischemic myocardium as soon as possible to reduce infarct size and associated complications. A recent pilot-study showed a significant reduction in infarct size by the induction of pre-reperfusion hypothermia.

Objectives: To demonstrate a reduction in infarct size/myocardium at risk (measured by magnet resonance imaging) in patients with ST-Elevation myocardial infarction by strategic temperature management with the use of external cooling pads in the out-of-hospital setting and the continuation with cold saline and central venous catheter cooling in hospital. In a parallel translational study, the molecular effects of rapid and early cooling on inflammatory processes at the culprit lesion site will be defined.

Methodology: Randomized, prospective, controlled trial Number of subjects: 120 patients (60 per group) Investigational medical device: EMCOOLS flex pad is an external cooling pad, that consists of multiple cooling cells filled with a patented cooling gel. EMCOOLS flex pad will be used in the out-of-hospital setting to initiate cooling. The Philips RTx Endovascular System™ is an endovascular thermal control system that circulates cooled saline through an indwelling central venous catheter in a closed-loop manner. It will be used in combination with 1-2 litres of intravenous cold saline to induce hypothermia below 35 degrees Celsius.

Duration: One hour after successful revascularization the cooling procedure will be stopped, subjects will be covered with a blanket and are allowed to passively re-warm. Clinical follow-up for 180 days.

Primary endpoint: Myocardial infarct size (as a percentage of myocardium at risk) assessed by cardiac MRI at 4±2 days. Influence of target temperature management on coronary macrophages and monocytes as well as impact on plasma levels of immune cell chemotaxis and activation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Immediate transfer to cath-lab is possible
* Anterior or inferior ST-segment myocardial infarction
* ST-Segment elevation of >0.2mV in 2 or more anatomically contiguous leads
* Duration of symptoms <6 hours

Exclusion Criteria:

* Participation in another study
* Patients presenting with cardiac arrest/cardiogenic shock
* Tympanic temperature <35.0°C prior to enrolment
* Thrombolytic therapy
* Previous MI
* Previous PCI or coronary artery bypass graft
* Severe heart failure at presentation (defined as a New York Heart Association (NYHA) functional class III or IV), or Killip classes II through IV
* Clinical signs of active infection
* End-stage kidney disease or hepatic failure
* Recent stroke (within the past six months)
* Conditions that may be exacerbated by hypothermia, such as haematological dyscrasias, oral anticoagulant treatment with international normalized ratio >1.5, severe pulmonary disease
* Pregnancy
* Women of childbearing potential
* Allergy to meperidine, buspirone, magnesium, or polyvinyl chloride
* Use of a monoamine oxidase inhibitor such as selegiline in the previous 14 days
* absolute contraindications against MRI (PM, ICD, ferromagnetic implants)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-02; Primary Completion 2016-07 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Infarct size (as percentage of myocardium at risk) assessed by cardiac MRI | Day 4±2
  The primary objective of this study is to demonstrate a reduction in infarct size (as percentage of myocardium at risk) assessed by cardiac MRI at 4±2 days when ST-elevation myocardial infarction is treated with primary coronary intervention (PCI) plus hypothermia compared to PCI alone

SECONDARY OUTCOMES:
Incidence of major adverse cardiac events | 6 months
  The effect of the hypothermia protocol on the incidence of the composite of death, heart failure, recurrent MI, malignant arrhythmias (i.e. ventricular fibrillation, sustained ventricular tachycardia) emergent stent revascularisation or any hospitalisation at 45±15 days and 6 months.
Immune cell activation | 4±2 days
  Impact of hypothermia on the number, the activation state, the adhesion and transmigratory capacity of coronary and systemic neutrophils and monocytes as well as impact of hypothermia on coronary and systemic plasma levels of soluble proteins related to innate immune cell chemotaxis and activation.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Testori, MD, Principal Investigator — Medical University of Vienna, Dept. of Emergency Medicine
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Mangold A, Ondracek AS, Hofbauer TM, Scherz T, Artner T, Panagiotides N, Beitzke D, Ruzicka G, Nistler S, Wohlschlager-Krenn E, Winker R, Quehenberger P, Traxler-Weidenauer D, Spannbauer A, Gyongyosi M, Testori C, Lang IM. Culprit site extracellular DNA and microvascular obstruction in ST-elevation myocardial infarction. Cardiovasc Res. 2022 Jun 29;118(8):2006-2017. doi: 10.1093/cvr/cvab217. PMID 34173822
- [Derived] Testori C, Beitzke D, Mangold A, Sterz F, Loewe C, Weiser C, Scherz T, Herkner H, Lang I. Out-of-hospital initiation of hypothermia in ST-segment elevation myocardial infarction: a randomised trial. Heart. 2019 Apr;105(7):531-537. doi: 10.1136/heartjnl-2018-313705. Epub 2018 Oct 25. PMID 30361270